CLINICAL TRIAL: NCT01105988
Title: A Pilot Study to Evaluate Tumor Pseudoprogression With FLT-PET and MRI
Brief Title: Evaluating Tumor Pseudoprogression With FLT-PET and MRI
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Funding ended
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Elizabeth R. Gerstner, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-008
Record Dates: First submitted 2010-04-15; First posted 2010-04-19 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Glioblastoma
Keywords: GBM; PET scans; MRI scans
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Radiologic exams — FLT PET scan x 2 MRI scan x 2

SUMMARY:
A standard treatment for glioblastoma is a combination of radiation and the drug temozolomide. This combination sometimes causing swelling (inflammation) of the brain tissue. When standard monitoring with MRI or CT scans is done within a few months of finishing treatment, it may be hard to tell if the scans are showing post-treatment brain inflammation or tumor growth and worsening of disease. Currently the only way to definitively distinguish inflammation from tumor growth is biopsy.

However, biopsy is an invasive procedure that is associated with risks. Having a non-invasive method to distinguish post-treatment inflammation from tumor growth can help improve care for patients with glioma.

For the PET scans in this research study, the investigators are using a radioactive substance called FLT (3'-deoxy-3'-[F-18] fluorothymidine), instead of the standard substance FDG (fluorodeoxyglucose). FLT gets absorbed by cancer cells but not by areas of inflammation. Because of that FLT may be better than FDG in differentiating cancer cells from inflammation.

An MRI scan will also be done at the same time as each of the 2 FLT-PET scans done for this research study. The two MRI scans performed will also help give more information about the patient's tumor that is not routinely provided with a routine clinical scan, such as blood flow through the tumor or metabolic activity in the tumor. The information from these special MRI scans may provide more information about the blood supply to the tumor and how this changes in response to treatment. In addition, the MRI scans along with the FLT-PET scans may help how to distinguish inflammation due to radiation therapy from tumor growth.

DETAILED DESCRIPTION:
If you are eligible to participate in this study you will have a pre-treatment FLT-PET scan within 7 days before starting treatment with radiation and temozolomide.

Two intravenous catheters (IVs) will be placed for each scan. One IV will be used to inject the FLT for the PET scan and the contrast agent for the MRI scan. The second IV will be used to draw blood for research tests. The PET scan will take about 2 hours. The MRI scan will take about 60-75 minutes. They will be done simultaneously.

About 4 weeks after you finish radiation therapy you will have a second FLT-PET scan and MRI scan.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed newly diagnosed glioblastoma
* Planned treatment for glioblastoma is standard radiation and temozolomide
* Measurable disease
* Life expectancy >/= 12 weeks
* Lab values must be within limits specified in protocol
* Able to undergo MRI and PET scans
* On stable dose of steroids for 5 days prior to each MRI scan

Exclusion Criteria:

* Chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering study or not recovered from adverse events from prior therapy
* Receiving any other study agents to treat tumor
* History of allergic reactions to compounds of similar chemical or biologic composition to FLT
* Uncontrolled intercurrent illness
* Pregnant or nursing
* HIV-positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure | 2 years
  To determine if elevated FLT PET uptake 4 weeks after completion of chemoradiation is associated with early tumor growth rather than treatment effect in patients with newly diagnosed glioblastome treated with standard chemoradiation.

SECONDARY OUTCOMES:
Secondary Outcome Measure | 2 years
  To clarify the impact of radiation and temozolomide chemotherapy on tumor cell proliferation.
Secondary Outcome Measure | 2 years
  To compare blood-derived kinetic parameters of tumor cell proliferation rate with image derived parameters of proliferation.
Secondary Outcome Measure | 2 years
  To examine the association of FLT uptake and MRI parameters, specifically contrast enhancement, perfusion, permeability, diffusion, and MR Spectroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Gerstner, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States